CLINICAL TRIAL: NCT05940337
Title: FIT to Grow Old - Functionality of the Immune System and Healthy Aging
Acronym: FTGO
Status: Completed | Type: Observational
Sponsor: Wageningen University (Other)
Collaborators: Top Consortium for Knowledge and Innovation (TKI) Argi & Food (Unknown); Mead Johnson Nutrition (Industry); Hycult Biotech (Unknown)
Responsible Party: Principal Investigator, Lydia A. Afman, Associate professor, Wageningen University
Other Study IDs: NL70696.081.19
Record Dates: First submitted 2022-07-01; First posted 2023-07-11 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Aging
Keywords: Immunometabolism; Monocyte; Elderly; Immune cell fitness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples are used to obtain circulating monocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elderly
- Young adults

SUMMARY:
Aging is commonly associated with reduced functionality of the immune system, resulting in a higher prevalence of infectious disease, auto-immune disease, cancer, and lower efficiency of vaccination. Nutritional strategies are increasingly recognized as a method to improve immune functionality, as several nutrients are shown to exert immunomodulatory properties. However, the large variation between individuals with regard to immune responses asks for more personalized approaches. Therefore, this field of research would benefit from a selection of those individuals with immune dysfunction. It is recently shown that immune functionality is largely dependent on intracellular metabolism, leading to the introduction of the new term 'immune cell fitness' which combines the metabolic and functional status of an immune cell. Within this study, we will determine the immune cell fitness of monocytes from healthy young adults and elderly subjects by measuring and integrating a broad range of metabolic and functional immune parameters into an immune cell fitness score. We aim to identify those individuals with immune dysfunction, the unfit. Furthermore, to identify potential nutritional strategies to improve immune cell fitness, we will study the effects of metabolites and nutrients on the immune cell fitness status of monocytes from elderly subjects.

DETAILED DESCRIPTION:
Rationale: Aging is commonly associated with reduced functionality of the immune system, resulting in a higher prevalence of infectious disease, auto-immune disease, cancer, and low-er efficiency of vaccination. The reduction in immune functionality is called 'immunosenescence' and is often observed in addition to a chronic state of systemic inflammation, referred to as 'inflammaging'. It is commonly believed that strategies improving immune functionality can be applied to improve healthy aging. Nutritional strategies, in particular, receive increasing attention, as several foods and nutrients are shown to exert immunomodulatory properties. Nutritional strategies focussing on the intake of polyunsaturated fatty acids have indeed shown improvements in cytokine profiles and inflammatory gene expression, but suffer from large inter-individual variation, which might be caused by differences in immune functionality. Recent studies within the field of immunometabolism have shown that immune functionality is largely dependent on intracellular metabolism, leading to the introduction of the new term ' immune cell fitness' which combines the metabolic and functional status of an immune cell. To improve the efficiency of immunomodulatory nutritional intervention strategies and work towards personalized approaches to support healthy aging, identifying individuals with reduced immune cell fitness will be crucial.

Objective: The primary aim of this study is to extensively characterize immune cell fitness in the elderly population to distinguish immunologically fit elderly from the unfit. Since immune cell fitness is a new concept, we will define a good immune cell fitness state using a young adult study population. Using a follow-up visit, we will evaluate whether our measure of immune cell fitness is robust and stable over time. Furthermore, to identify potential nutritional strategies to improve immune cell fitness and work towards personalized approaches, we will study the effects of metabolites and nutrients on their ability to improve immune cell fitness in monocytes from the elderly.

Study design: The study will be a cross-sectional study in which we will compare the immune cell fitness state of elderly people using young adult people to define an 'immune fit' status. Immune cell fit-ness will be measured in monocytes, which will be obtained from blood samples. Subjects will be given a standardized meal which they consume in the evening before the study visit at latest 8.00 pm. After consumption of the meal, subjects are not allowed to eat or drink anything but water.

On the study day, before the start of blood sampling, a small blood sample via a finger prick is collected to measure CRP levels. CRP levels of ≥10.0 mg/L indicate severe infection and will consequently exclude the subject from participating on that specific day. The relevant subjects are asked to make a new appointment. If CRP levels are < 10 mg/L, blood sampling will continue.

Blood sampling and anthropometric measurements including body weight, waist and hip circumference and a DEXA scan will be performed in each subject, after which the subjects will receive breakfast. Subjects will fill in an FFQ to gain insights into regular dietary intake. In addition, subjects will fill in questionnaires on sleep quality and general health.

Elderly subjects will be contacted for a follow-up visit at least 6 months and the latest 18 months after the study visit. The study-design of the follow-up visit will be similar to the first study visit, including the standardized meal the evening before, overnight fast, blood sampling, anthropometric measurements (except for the DEXA-scan, this will only be performed as a link between immune cell fitness and fat distribution is found in the first part of the study), and questionnaires. The freshly collected blood sample will be used for our secondary aims, namely 1) to study the effects of nutrients and metabolites on immune cell fitness, and 2) to test whether our measure of immune cell fitness is robust and stable over time.

Update August 2023 Based on our preliminary results, we decided to cancel the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 30y and 60 - 75y
* BMI 18.5 - 25 kg/m2 (young adults); 20 - 30 kg/m2 (elderly)
* Willing to fast overnight for 12 hours
* Willing to give a blood sample
* Having a general practitioner
* Signed informed consent

Exclusion Criteria:

* Diagnosed with metabolic and/or inflammatory disease (e.g. diabetes, cardiovascular disease (with the exception of hypertension), arthritis, arthrosis, glycogen storage dis-orders and auto-immune diseases)
* Current diagnosis of cancer
* Regular use of medication that interferes with immune function (e.g. corticosteroids, cytokine blockers)
* Regular use of medication that may interfere with metabolism (e.g. metabolic inhibitors or activators)
* Use of medication that interferes with immune function and metabolism in at least one week preceding the study visit (e.g. NSAID, anti-histamines, corticosteroids)
* More than 4kg weight gain or weight loss over the last 4 months
* Vaccination within 3 months preceding the study visit (e.g. immunization against influ-enza, pneumonia, and travel-related infections)
* Donated blood within 2 months preceding the study visit
* Pregnant, lactating or wishing to become pregnant in the period between the screening and study visit (self-reported)
* Regular use of hard drugs and soft drugs (i.e. weekly use) and at least no use within 2 months preceding the study visit
* Excessive alcohol use (i.e. >14 units per week)
* Use of cigarettes and other tobacco products
* Participation in another study that involves an intervention 2 months preceding the study visit
* Members of the research team
* Working, or doing an internship or thesis at the division "Human Nutrition and Health", Wageningen University

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of healthy men and women between the age of 20 - 30 years old and between 60 - 75 years old. The ratio between men and women will be kept equally as much as possible in both groups. The young adults should have a BMI between 18.5 - 25 kg/m2. The elderly subject should have a BMI between 20 - 30 kg/m2. Subjects will be recruited from the surroundings of Wageningen using the mailing list for potential research subjects from the division of Human Nutrition and Health, Wageningen University.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Lactate production | 1 day
  Lactate excretion by monocytes after ex-vivo exposure to inflammatory stimuli
Cytokine production | 1 day
  Cytokine excretion by monocytes after ex-vivo exposure to inflammatory stimuli. Measured using ELISA for IL-6, IL-1b. IL-1RA, IL-8, TNFalpha.

SECONDARY OUTCOMES:
Phagocytosis | 1 day
  Phagocytic capacity of monocytes. Measured using absorbed fluorescent beads and flow cytometry.
Glycolytic and oxidative capacity | 1 day
  Glycolytic and oxidative capacity of monocytes. Measured using Seahorse Assays (Agilent).

OTHER OUTCOMES:
Circulating immune mediators | 1 day
  Circulating cytokines and other immune related markers in plasma
Glucose levels | 1 day
  circulating glucose concentration in plasma
Lipid profile | 1 day
  Circulating lipids (Triglycerides, HDL and LDL)
Anthropometric measures - body weight | 1 day
  Bodyweight in kg
Anthropometric measures - body height | 1 day
  bodyheight in cm
Anthropometric measures - WHR | 1 day
  waist- and hip-circumference in cm
Anthropometric measures - DEXA | 1 day
  Dual Energy Xray absorptiometry to measure fat distribution in percentages of total mass, total body
C-reactive protein | 1 day
  Concentrations in whole blood and plasma
Questionnaires - FFQ | 1 day
  Food frequency questionnaire. Results are expressed as the average amount of portions consumed weekly for each food group (e.g. bread, spread, snacks, cold meal, warm meal).
Questionnaires - general health | 1 day
  General health questionnaires. Questionnaires are translated into Dutch and therefore not validated. Answers will be coded and used for analysis. Some questions include a score from 1 to 5 or 10, where low scores represent bad outcomes or not frequent, and high scores represent good outcomes or frequent.
Questionnaires - sleep quality | 1 day
  Sleep quality questionnaires. Questionnaires are translated into Dutch and therefore not validated. Answers will be coded and used for analysis. Some questions include a score from 1 to 5 or 10, where low scores represent bad outcomes or not frequent, and high scores represent good outcomes or frequent.
Gene expression | 1 day
  expression of metabolic and inflammatory genes in monocytes and macrophages at baseline and after stimulation with pro-inflammatory mediators. Measured using qPCR and RNAsequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Afman, Principal Investigator — Wageningen University; Rinke Stienstra, Principal Investigator — Wageningen University
Locations (1):
- Department of Human Nutrition & Health, Wageningen University, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
All research subjects will get a numeric code (Pxx-Pxx) that is coupled to their personal data. Personal data will be stored in a closed locker and a password-protected file. Only the investi-gators will have access to the key of the code. The same code will also be used to code the collected material. Subsiding partners do not have access to personal data or material. This will all be done in line with the General Data Protection Regulation (GDPR) effective from the 25th of May 2018 onwards.

REFERENCES:
- [Derived] Smeehuijzen L, Vrieling F, Jansen J, van der Zande HJP, Houslay TM, Gross G, van Diepen JA, Afman LA, Stienstra R. Lactate Secretion by Monocytes as a Determinant of Innate Immune Cell Fitness in Healthy Elderly. Aging Cell. 2025 Nov;24(11):e70220. doi: 10.1111/acel.70220. Epub 2025 Oct 13. PMID 41078099